CLINICAL TRIAL: NCT00541333
Title: Weekly Vaccination With Copaxone as a Potential Therapy for Dry Age-related Macular Degeneration
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Reviewing data
Sponsor: The New York Eye & Ear Infirmary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NYEE100907
Record Dates: First submitted 2007-10-09; First posted 2007-10-10 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Dry Age Related Macular Degeneration
Keywords: Dry Age Related Macular Degeneration; Dry AMD
MeSH Terms: interventions — Glatiramer Acetate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Copaxone (Active Comparator)
  Interventions: Drug: Copaxone Injection
- Sham (Sham Comparator)
  Interventions: Drug: Copaxone Injection

INTERVENTIONS:
Drug: Copaxone Injection

SUMMARY:
The purpose of the project is to investigate in eyes with dry AMD, the efficacy and safety as preventive therapy of the immunomodulatory substance named copaxone which had been proven as safe and effective agent for a neurodegenerative disease, in arresting the progression as well as the conversion of dry AMD to wet AMD. The hypothesis that the immunomodulatory agent copaxone proven for a neurodegenerative disease may work in the eye is revolutionary and may open a new avenue of preventive treatment for the disease which is the major cause of legal blindness in the industrial world

ELIGIBILITY:
Inclusion Criteria:

1. Dry AMD in one or both eyes
2. Age 50 or above of either gender
3. Signed informed consent.

Exclusion Criteria:

1. Known sensitivity to Mannitol or Copaxone.
2. Skin disease or active infection of skin.
3. Active fever or active treatment for infection.
4. History of other uncontrolled systemic active disease.
5. Premenopausal females not using reliable birth control.
6. Sensitivity to fluorescein or iodine.
7. Inability to comply with study procedures.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-12; Primary Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Total drusen area reduction | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Richard B Rosen, MD, Principal Investigator — New York Eye and Ear Infirmary
Locations (1):
- New York Eye and Ear Infirmary, New York, New York, United States